CLINICAL TRIAL: NCT00004010
Title: Pilot Study for the Treatment of Children With Newly Diagnosed Advanced Stage Hodgkin's Disease: Upfront Dose Intensive Chemotherapy
Brief Title: Combination Chemotherapy and Radiation Therapy in Treating Children With Previously Untreated Stage II, Stage III, or Stage IV Hodgkin's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 59704; COG-59704 (Other: Children's Oncology Group); CDR0000067222 (Other: ClinicalTrials.gov)
Record Dates: First submitted 1999-11-01; First posted 2004-04-15 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Lymphoma
Keywords: stage II childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; childhood lymphocyte predominant Hodgkin lymphoma; childhood lymphocyte depletion Hodgkin lymphoma; childhood nodular sclerosis Hodgkin lymphoma; childhood mixed cellularity Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Bleomycin; Filgrastim; ABVD protocol; Cyclophosphamide; Dacarbazine; Doxorubicin; Etoposide; Prednisone; Procarbazine; Vinblastine; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BEACOPP therapy (Experimental): Patients receive 4 cycles of BEACOPP therapy. Drugs utilized in this regimen include Bleomycin (B), Etoposide (E), Doxorubicin (A), Cyclophosphamide (C), Vincristine (O), Prednisone (P) and Procarbazine (P). Each cycle lasts 21 days and is characterized by intravenous pulses of Etoposide (Days 0-2), Doxorubicin (Day 0), Cyclophosphamide (Day 0), Bleomycin (Day 7), Vincristine (Day 7). Seven days of oral procarbazine (Days 0-6) and 14 days of oral prednisone (Days 0-13) are given during each cycle.
  Growth factor support with Filgrastim (G-CSF) is given by subcutaneous injection daily beginning Day 8. Response will then be determined and stratification for further treatment.
  Interventions: Biological: bleomycin sulfate; Biological: filgrastim; Drug: ABVD regimen; Drug: cyclophosphamide; Drug: dacarbazine; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: prednisone; Drug: procarbazine hydrochloride; Drug: vinblastine sulfate; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Biological: bleomycin sulfate
  Other Names: Blenoxane
Biological: filgrastim
  Other Names: GCSF; Neupogen
Drug: ABVD regimen
Drug: cyclophosphamide
  Other Names: Cytoxan
Drug: dacarbazine
Drug: doxorubicin hydrochloride
  Other Names: Adriamycin
Drug: etoposide
  Other Names: VP-16; VePesid
Drug: prednisone
Drug: procarbazine hydrochloride
  Other Names: Matulane
Drug: vinblastine sulfate
  Other Names: Velban
Drug: vincristine sulfate
  Other Names: Oncovin; Vincasar; VCR; leurocristine; NSC# 67574
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. Radiation therapy uses high-energy x-rays to damage cancer cells. Giving radiation therapy after chemotherapy may be an effective treatment for Hodgkin's disease.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy and radiation therapy in treating children who have previously untreated stage II, stage III, or stage IV Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility and toxicity of bleomycin, etoposide, doxorubicin, cyclophosphamide, vincristine, procarbazine, and prednisone (BEACOPP) induction in pediatric patients with previously untreated stage II, stage III, or stage IV Hodgkin's disease. II. Determine rates of complete response and rapid early partial response (defined as greater than 70% reduction in the size of a bulky mediastinal mass or nodal aggregate and a negative gallium scan) in these patients treated with 4 courses of BEACOPP. III. Determine whether thallium scans effectively measure response to therapy in these patients treated with this regimen. IV. Evaluate the expression of markers of apoptosis in tumor samples from these patients at diagnosis and at time of relapse, and correlate expression of these markers with response to therapy and overall outcome. V. Determine the utility of seven molecular genetic markers as surrogate markers of genotoxic damage caused by this regimen in these patients. VI. Estimate the incidence of therapy related late effects, including second malignant neoplasms, sterility, cardiac dysfunction, pulmonary restrictive disease, growth abnormalities, and thyroid disease in these patients.

OUTLINE: Induction: On day 0, patients receive cyclophosphamide IV over 30 minutes, doxorubicin IV over 15-30 minutes, etoposide IV over 1 hour, oral prednisone every 12 hours, and oral procarbazine. On days 1 and 2, patients receive etoposide IV over 1 hour, oral prednisone every 12 hours, and oral procarbazine. On days 3-6, patients receive oral prednisone every 12 hours and oral procarbazine. On day 7, patients receive vincristine IV, bleomycin IV over 5 minutes, and oral prednisone every 12 hours. On days 8-13, patients receive oral prednisone every 12 hours. Beginning on day 8, patients receive filgrastim (G-CSF) subcutaneously until absolute neutrophil counts recover. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Consolidation therapy begins on week 12 or when blood counts recover. Consolidation for rapid early responders (patients with complete response (CR) or rapid early partial response (PR-1) to induction therapy): Females - Patients receive vincristine IV, cyclophosphamide IV over 30 minutes, oral prednisone every 12 hours, and oral procarbazine on day 0. On days 1-6, patients receive oral prednisone every 12 hours and oral procarbazine. On day 7, patients receive vinblastine IV, bleomycin IV over 5 minutes, doxorubicin IV over 15-30 minutes, and oral prednisone every 12 hours. On days 8-13, patients receive oral prednisone every 12 hours. Treatment repeats every 28 days for a total of 4 courses in the absence of disease progression or unacceptable toxicity. Males - Patients receive doxorubicin IV over 15-30 minutes, bleomycin IV over 5 minutes, vinblastine IV, and dacarbazine IV on days 0 and 14. Treatment repeats every 28 days for a total of 2 courses in the absence of disease progression or unacceptable toxicity. Beginning 3 weeks after completion of chemotherapy, male patients with CR or PR-1 receive radiotherapy 5 days per week to areas of initial disease involvement (total duration of radiotherapy is dependent on initial extent of disease). Consolidation for slow early responders: Patients with slow partial response (PR-2) or stable disease (SD) after 4 courses of induction therapy receive 4 additional courses of induction therapy in the absence of disease progression or unacceptable toxicity. Beginning on day 8, patients receive G-CSF subcutaneously until blood counts recover. Patients should be off G-CSF for more than 24 hours prior to the next course of chemotherapy. Beginning 3 weeks after completion of chemotherapy, male and female patients with PR-2 or SD receive radiotherapy 5 days per week to areas of initial disease involvement (total duration of radiotherapy is dependent on initial extent of disease). Patients are followed every 3 months for 2 years, every 6 months for 1 year, annually for 2 years and then at years 10 and 20.

PROJECTED ACCRUAL: Approximately 25-50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven, previously untreated Hodgkin's disease Stage IV OR Stage II or stage III with B symptoms (at least 1 of the following: unexplained weight loss greater than 10%, unexplained recurrent fever greater than 39 degrees C, or drenching night sweats) AND bulk disease (defined as a mediastinal mass greater than 1/3 of mediastinal thoracic diameter and/or nodal aggregate greater than 10.0 cm) The following cellular types are eligible: Mixed cellularity, not otherwise specified (NOS) Lymphocytic depletion, NOS Lymphocytic depletion, diffuse fibrosis Lymphocytic depletion, reticular Lymphocytic predominance, NOS Lymphocytic predominance, diffuse Lymphocytic predominance, nodular Hodgkin's paragranuloma Hodgkin's granuloma Hodgkin's sarcoma Nodular sclerosis, NOS Nodular sclerosis, cellular phase Nodular sclerosis, lymphocytic predominance Nodular sclerosis, mixed cellularity Nodular sclerosis, lymphocytic depletion Hodgkin's disease, NOS Must begin protocol therapy within 42 days of biopsy and 7 days of completion of staging

PATIENT CHARACTERISTICS: Age: 21 and under Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: No prior treatment for Hodgkin's disease

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 1999-10; Primary Completion 2003-10 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Estimate the rate of BEACOPP )((Bleomycin, Etoposide, Adriamycin, Cyclophosphamide, Vincristine, Procarbazine, Prednisone) specific toxicity in pediatric patients

SECONDARY OUTCOMES:
Obtain preliminary estimates of response to BEACOPP ((Bleomycin, Etoposide, Adriamycin, Cyclophosphamide, Vincristine, Procarbazine, Prednisone)

CONTACTS AND LOCATIONS:
Overall Officials: Kara Kelly, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (40):
- United States (37):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia

REFERENCES:
- [Result] Kelly KM, Sposto R, Hutchinson R, Massey V, McCarten K, Perkins S, Lones M, Villaluna D, Weiner M. BEACOPP chemotherapy is a highly effective regimen in children and adolescents with high-risk Hodgkin lymphoma: a report from the Children's Oncology Group. Blood. 2011 Mar 3;117(9):2596-603. doi: 10.1182/blood-2010-05-285379. Epub 2010 Nov 15. PMID 21079154
- [Result] Kelly M, Hutchinson R, Sposto R, et al.: BEACOPP chemotherapy is a highly effective regimen in children and adolescents with advanced stage Hodgkin's disease: results from Children's Cancer Group study CCG-59704. [Abstract] Eur J Haematol 75 (Suppl 65): A-WP07, 72, 2004.
- [Result] Shiramizu B, Morris E, Perkins S, et al.: Identification of patient specific primers (PSPs) of IgH and TCR-y regions by nested PCR in CD20 positive Hodgkin disease: a Children's Cancer Group report (CCG). [Abstract] Ann Oncol 13(suppl 2): A-389, 112, 2002.